CLINICAL TRIAL: NCT05166902
Title: Evaluation of Monthly Replacement Lens Designs in Habitual Soft Contact Lens Wearers Who Report Frequent Digital Devise Use
Brief Title: Evaluation of Monthly Replacement Lenses in Habitual Soft Contact Lens Wearers Who Report Frequent Digital Devise Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Collaborators: Centre for Ocular Research & Education, Canada (Other)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EX-MKTG-130
Record Dates: First submitted 2021-12-08; First posted 2021-12-22 (Actual); Results first posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2022-05

CONDITIONS: Ametropia
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Lens A, Then Lens B (Experimental): Participants will wear lens A for one month and then cross over to wear lens B for one month.
  Interventions: Device: Lens A (comfilcon A lens); Device: Lens B (lehfilcon A lens)
- Lens B, Then Lens A (Experimental): Participants will wear lens B for one month and then cross over to wear lens A for one month.
  Interventions: Device: Lens A (comfilcon A lens); Device: Lens B (lehfilcon A lens)

INTERVENTIONS:
Device: Lens A (comfilcon A lens) — 1 month
Device: Lens B (lehfilcon A lens) — 1 month

SUMMARY:
To evaluate the clinical performance of two monthly silicone hydrogel contact lenses in habitual wearers of frequent replacement (FRP) lenses when worn for 1-month.

DETAILED DESCRIPTION:
This study is a prospective, bilateral eye, double-masked, randomized, 1-month cross-over, daily-wear design involving two different FRP lens types. Each lens type will be worn for approximately one month.

ELIGIBILITY:
Inclusion Criteria:

1. Is at least 18 years of age and no older than 35 years, and has full legal capacity to volunteer;
2. Has read and signed an information consent letter;
3. Is willing and able to follow instructions and maintain the appointment schedule;
4. Self-reports having a full eye examination in the previous two years;
5. Self-reports spending on most days at least 6 hours cumulative (not necessarily in one single stretch) using digital devices such as a computer, laptop, tablet, e-reader, smartphone;
6. Has healthy eyes with no health condition or medication that contra-indicate contact lens wear, in the opinion of the investigator;
7. Anticipates being able to wear the study lenses for at least 8 hours a day, 6 days a week;
8. Habitually wears soft frequent replacement contact lenses, for the past 3 months minimum (NOTE: The habitual contact lens brand was restricted such that no more than one third were to be Biofinity Energys brand (or their equivalent private label brand name) and no more than one third were to be Alcon brand);
9. Has refractive astigmatism no higher than -0.75DC in each eye;
10. Can be fit and achieve binocular distance vision of at least 20/30 Snellen (Available lens parameters are sphere +6.00 to -6.00D, 0.25D steps).

Exclusion Criteria:

1. Is participating in any concurrent clinical or research study;
2. Has any known active ocular disease and/or infection that contraindicates contact lens wear;
3. Has a systemic or ocular condition that in the opinion of the investigator may affect a study outcome variable;
4. Is using any systemic or topical medications that in the opinion of the investigator may affect contact lens wear or a study outcome variable;
5. Has known sensitivity to the diagnostic sodium fluorescein used in the study;
6. Self-reports as pregnant, lactating or planning a pregnancy at the time of enrolment;
7. Has undergone refractive error surgery or intraocular surgery.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2022-07-09 (Actual); Study Completion 2022-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Wilkinson, Principal Investigator — Spadina Optometry; Roxanne Achong-Coan, Principal Investigator — Coan Eyecare; Fiona Soong, Principal Investigator — Eyes on Sheppard Clinic; Mike Cymbor, Principal Investigator — Nittany Eye Associates
Locations (4):
- United States (2):
  - Coan Eye Care, Ocoee, Florida
  - Nittany Eye Associate, State College, Pennsylvania
- Canada (2):
  - Eyes on Sheppard Clinic, Toronto, Ontario
  - Spadina Optometry, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Sixty-seven participants were screened with no screen failures. One participant discontinued and the remaining 66 all completed the study.
  All the participants who completed the study were included in the analysis. (Analysis population n=66)
Groups:
- Lens A, Then Lens B: Participants wore Lens A for one month and then crossed over to wear Lens B for one month.
- Lens B, Then Lens A: Participants wore Lens B for one month and then crossed over to wear Lens A for one month.
Period: First Intervention
Arm/Group | Lens A, Then Lens B | Lens B, Then Lens A
Started | 34 | 33
Completed | 34 | 32
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Second Intervention
Arm/Group | Lens A, Then Lens B | Lens B, Then Lens A
Started | 34 | 32
Completed | 34 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Sixty-six participants completed the study, and demographic data include all participants who completed the study.
Groups:
- Analysis Population: Sixty-six participants completed the study, and demographic data include all participants who completed the study.
Arm/Group | Analysis Population
Number analyzed (Participants) | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 66
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.8 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Subjective Ratings on Lens Handling on Removal
Description: Subjective ratings on lens handling on removal will be measured on a scale of 0-10, 0.5 steps (10= Very Easy, 0= Very Difficult)
Time Frame: Day 27
Population: Participants
Measure: Mean (Standard Deviation); unit: Units on scale
Groups:
- Lens A: Participants wore Lens A for 1 month.
- Lens B: Participants wore Lens B for 1 month.
Arm/Group | Lens A | Lens B
Number analyzed (Participants) | 66 | 66
Units on scale | 8.3 (1.8) | 8.8 (1.2)

ADVERSE EVENTS:
Time Frame: From dispense up to one month on each study lens, for total of two months
Description: [Not Specified]
Groups:
- Lens A: Participants wore Lens A for one month
- Lens B: Participants wore Lens B for one month
Arm/Group | Lens A | Lens B
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/66
Other Adverse Events (participants affected / at risk) | 4/66 | 2/66
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lens A (N=66) | Lens B (N=66)
COVID-19 (Social circumstances) | 3 | 1
Lens discomfort (Product Issues) | 1 | 0
Sinus (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/02/NCT05166902/Prot_SAP_000.pdf